CLINICAL TRIAL: NCT00301561
Title: Expanded Access to Antiretroviral Therapy in Africa: Assessment of the Patients' Management in District Hospitals With a Simplified Follow-up Approach (ANRS 12110 STRATALL)
Brief Title: Antiretroviral Treatment Simplified Follow-up Management Assessment (ANRS 12110 STRATALL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12110 STRATALL
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: HIV Infections; AIDS
Keywords: Antiretroviral treatment; Expanded access; Africa; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Simplify treatment follow-up
  Interventions: Procedure: Simplified follow-up approach of ARV treatment
- 2 (Active Comparator): Standard treatment follow-up
  Interventions: Procedure: Standard follow-up approach of ARV treatment

INTERVENTIONS:
Procedure: Simplified follow-up approach of ARV treatment — Simplify treatment follow-up :
  * some clinical consultations will be performed by nurses under the physicians' responsibility ;
  * the CD4 cell count and HIV-1 viral load will not be available for the management of patients ;
  * the biologic assessment for tolerability will be limited
  Arms: 1
Procedure: Standard follow-up approach of ARV treatment — Standard treatment follow-up :
  * all clinical consultations will be performed by physicians ;
  * the CD4 cell count and HIV-1 viral load will be available for the patients management routinely ;
  * the biologic assessment for tolerability will be available as needed
  Arms: 2

SUMMARY:
Access to antiretroviral therapy (ART) is still limited in Africa (11% of patients in immediate need in June 2005). Face to the scope of the need and the constraints (unavailability and cost of viral load and CD4 cell count, lack of physicians…), WHO has developed a follow-up approach based on a simplified monitoring. However, this "simplified" approach which represents a major stake for the expanded access to ART has been little evaluated against the gold standard approach.

DETAILED DESCRIPTION:
Justification

Access to antiretroviral therapy (ART) is still limited in Africa (11% of patients in immediate need in June 2005). Face to the scope of the need and the constraints (unavailability and cost of viral load and CD4 cell count, lack of physicians…), WHO has developed a follow-up approach based on a simplified monitoring. This "simplified" approach restricting the use of complementary exams including biologic criteria of effectiveness and tolerability, some people consider this approach as dangerous for the patient but also for the community (rapid emergence of resistances) and that it would be preferable to treat less patients and only with the gold standard approach. In practice, this "simplified" approach which represents a major stake for the expanded access to ART has been little evaluated against the gold standard approach.

Objectives

Main objective: To compare the increase in the CD4 cell count in patients receiving ART with a "simplified" approach and in those treated with the gold standard approach in district hospitals.

Secondary objectives: To compare between the two approaches the virologic effectiveness, survival, treatment interruptions, number of patients lost to follow-up, clinical progression, clinical and biologic tolerability, adherence, emergence of drug resistances, impact on patients' daily life, acceptability by the patients and health professionals, and cost-effectiveness performances.

Methods

Randomised, controlled, multicentre, non inferiority, intervention trial, without blind for approach, in 9 district hospitals of the Province du Centre in Cameroon. 430 adult patients will be randomised in two groups ("simplified" approach or gold standard approach) with a 1:1 ratio and followed for 24 months.

In the "simplified" approach, the results of the HIV-1 viral load and CD4 cell count will not be available for the management of patients, the biologic assessment of tolerability will be limited and some clinical consultations will be performed by nurses under the physicians' responsibility; the remainder will be similar to the gold standard approach.

Planning

The study will start in the first semester of 2006. The full length of the study would be 36 months maximum (12 months for enrolment and 24 months for follow-up).

Expected results

Advices for increasing access to ART in Africa.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged at least 18 years
* Living in the health district of the hospital attended
* Confirmed HIV-1 group M infection
* Meeting one of the following criteria:

  * Stage III or IV (WHO classification)
  * Stage II (WHO classification) and total lymphocytes count ≤ 1200/mm3
* Patient agreeing on monthly follow-up and treatment for 24 months
* Signed informed consent

Exclusion Criteria:

* HIV-1 group O or N, or HIV-2 infection
* HIV-1 primary infection
* Progressive tuberculosis in treatment and total lymphocytes count > 1200/mm3
* Progressive tumor or malignant lymphoma (except cutaneous or mucous Kaposi sarcoma)
* Progressive psychiatric disorder
* Hepatocellular disorder
* History of antiretroviral therapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2006-05; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Increase in the CD4 cell count measured with a FACSCount apparatus after 24 months of antiretroviral therapy | 24 months

SECONDARY OUTCOMES:
Percentage of patients with viral load below 400 copies/ml and 50 copies/ml, respectively (Abbott RealTime HIV-1) | 12 and 24 months
Survival probability | Through out the trial
Probability of treatment interruption | Through out the trial
Probability of patients lost to follow-up | Through out the trial
Incidence of side effects | Through out the trial
Incidence of clinical events (WHO stage III or IV) | Through out the trial
Percentage of adherence | 12 and 24 months
Percentage of patients with drug resistance | 12 and 24 months
Acceptability by the patients and health professionals of both approaches | 12 and 24 months
Impact on patients' daily life | Through out the trial
Cost-effectiveness ratio | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Laurent, Study Chair — Institut de Recherche pour le Developpement; Eric Delaporte, Study Chair — Institut de Recherche pour le Developpement; Sinata Koulla-Shiro, Study Chair — Hôpital Central, Yaoundé, Cameroun; Charles Kouandack, Study Chair — Hôpital Central, Yaoundé, Cameroun
Locations (9):
- Cameroon (9):
  - Hôpital de district d'Ayos, Ayos
  - Hôpital de district de Bafia, Bafia
  - Hôpital de district de Mfou, Mfou
  - Hôpital de district de Monatélé, Monatélé
  - Hôpital de district de Nanga Eboko, Naga Eboko
  - Hôpital de district de Ndikiniméki, Ndikiniméki
  - Hôpital de district d'Obala, Obala
  - Hôpital de district de Sa'a, Sa'a
  - Hôpital de district de Mbalmayo, Yaoundé

REFERENCES:
- [Derived] Sandie AB, Molinari N, Wanjoya A, Kouanfack C, Laurent C, Tchatchueng-Mbougua JB. Non-inferiority test for a continuous variable with a flexible margin in an active controlled trial: an application to the "Stratall ANRS 12110 / ESTHER" trial. Trials. 2022 Mar 5;23(1):202. doi: 10.1186/s13063-022-06118-x. PMID 35248123
- [Derived] Laurent C, Kouanfack C, Laborde-Balen G, Aghokeng AF, Mbougua JBT, Boyer S, Carrieri MP, Mben JM, Dontsop M, Kaze S, Molinari N, Bourgeois A, Mpoudi-Ngole E, Spire B, Koulla-Shiro S, Delaporte E; Stratall ANRS 12110/ESTHER study group. Monitoring of HIV viral loads, CD4 cell counts, and clinical assessments versus clinical monitoring alone for antiretroviral therapy in rural district hospitals in Cameroon (Stratall ANRS 12110/ESTHER): a randomised non-inferiority trial. Lancet Infect Dis. 2011 Nov;11(11):825-833. doi: 10.1016/S1473-3099(11)70168-2. Epub 2011 Aug 8. PMID 21831714